CLINICAL TRIAL: NCT02534571
Title: Endoscopic Application of a Hemostatic Powder TC-325 Versus Standard Treatment in the Control of Acute Upper Gastrointestinal Bleeding From Nonvariceal Causes; A Non-inferiority Randomized Trial
Brief Title: To Compare a Hemostatic Powder TC-325 and Standard Treatment in the Control of Acute Upper Gastrointestinal Bleeding From Nonvariceal Causes
Acronym: TC325
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Collaborators: North District Hospital (Other); King Chulalongkorn Memorial Hospital (Other); Changi General Hospital (Other)
Responsible Party: Principal Investigator, James Yun-wong Lau, Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TC325 Study
Record Dates: First submitted 2015-08-06; First posted 2015-08-27 (Estimated); Last update posted 2019-10-11 (Actual); Status verified 2019-10

CONDITIONS: Acute Upper Gastrointestinal Bleeding
MeSH Terms: interventions — Epinephrine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- TC-325 (Experimental): Endoscopic Application of a Hemostatic Powder TC-325, <=150gm , once
  Interventions: Device: Endoscopic Application of a Hemostatic Powder TC-325
- standard treatment (Active Comparator): standard treatment of either hemo-clipping or thermo-coagulation with or without pre injection with diluted epinephrine <=20 clip or4 pulse , once only
  Interventions: Device: Hemo-clipping; Drug: Epinephrine; Device: thermo-coagulation

INTERVENTIONS:
Device: Endoscopic Application of a Hemostatic Powder TC-325 — Endoscopic Application of a Hemostatic Powder TC-325 <=150g once
  Arms: TC-325
Device: Hemo-clipping — Hemo-clipping <=20 clips
  Other Names: quick clips
  Arms: standard treatment
Drug: Epinephrine — epinephrine injection endoscopically <20 mls
  Other Names: adrenaline
  Arms: standard treatment
Device: thermo-coagulation — contact thermo-coagulation < = 4 pulses
  Other Names: contact thermo-coagulation
  Arms: standard treatment

SUMMARY:
Acute upper gastrointestinal bleeding is a common medical emergency. Bleeding peptic ulcers and other non-variceal causes constitute to about 95% of all cases of bleeding. Endoscopic treatment stops active bleeding, reduces rate of further bleeding and leads to improved patients outcomes. Endoscopic treatment can be technically demanding especially with lesions in difficult anatomic positions and to endoscopists with less experience. TC-325 is a propriety mineral blend hemostatic powder used to compress external civilian and military traumatic injuries. Investigators reported the first endoscopic application of TC-325 in 20 patients with actively bleeding gastro-duodenal ulcers. Investigators were able to stop bleeding in 19 of them. Subsequent case series from others reported a similar rate in the acute control of bleeding. To further define the role of TC-325 as a mono-therapy, a comparison to the current standard in endoscopic treatment is required. A non-inferiority randomized trial is being proposed to compare endoscopic use of TC-325 as a mono-therapy to current standards (i.e. hemoclips or thermo-coagulation with or without pre-injection with diluted epinephrine) in hemostatic treatment in patients with acute upper gastrointestinal bleeding from non-variceal causes. The non-inferiority primary endpoint is control of bleeding over 30 days from randomization. Other outcome endpoints include further endoscopic, angiographic or surgical treatments, hospitalization, blood transfusion and mortality. Investigators also compare ease of therapy measured by procedure time and a 10 cm visual analogue scale rated by endoscopists. Endoscopic application of TC-325 is a simple and less skill dependent technique. It may prove useful in bleeding from anatomically challenging sites of the gastro-duodenal tract.

DETAILED DESCRIPTION:
Impact and Objectives Long-term impact :Acute upper gastrointestinal bleeding is a common medical emergency. The majority of causes are non-variceal in etiology and are mostly peptic ulcers. Endoscopic treatment reduces further bleeding, surgery and deaths from the condition. The current endoscopic treatment to non-variceal causes includes.the use of hemo-clips and thermo-coagulation. Endoscopic treatment is skill demanding and can be challenging in difficult access areas in the gastroduodenal tract e.g. posterior bulbar duodenum. Endoscopic application of hemostatic powder (labeled TC-325) is technically easy. The proposed randomized trial is the first to compare TC-325 to standard treatment. An non-inferior treatment of hemostatic powder TC-325 would mean wider application of endoscopic treatment as most endoscopists are able to use it. It can at least be used for acute control of bleeding allowing time for more definitive treatment.

Objectives :

1. To compare clinical efficacy of the hemostatic powder TC-325 to standard treatment in overall rate of hemostasis in patients with active bleeding from a non-variceal source in the upper gastrointestinal tract. Investigators aim to determine the initial rate of hemostasis and the rate of further bleeding after initial control in both groups. Investigators would like to define role of TC-325 as a mono-therapy when compared to standard treatment. The rate of further bleeding after initial control would also inform us if endoscopic application of TC-325 should be followed by a second look endoscopy with targeted treatment to the bleeding artery.
2. To compare ease of application of hemostatic powder TC-325 to standard treatment.

Background of Research, Research Plan and Methodology :

a. Background of research Acute upper gastrointestinal bleeding (AUGIB) is one of the commonest medical emergencies. Mortality in patients with AUGIB remains high. In the National United Kingdom Audit of 2007, the crude overall in patient mortality was 10%. Mortality increases in patients with advanced age and significant comorbid illnesses. Endoscopic therapy greatly improves outcomes in patients with AUGIB. In pooled analyses of randomized controlled trials on endoscopic therapy in patients with nonvariceal upper gastrointestinal bleeding, endoscopic therapy significantly reduces not only further bleeding but also surgery and deaths.

The National United Kingdom audit in 2007 found continuing delays in endoscopy and treatment in patients admitted with AUGIB. Only 55% of patients judged to belong to the high risk group underwent endoscopy within 24 hours of their admissions, and only 74% of high risk lesions were offered endoscopic treatment. The gap in service provision may be an organization issue. The lack of skills in endoscopic therapy may also contribute to this shortfall. An easy-to-use endoscopic treatment is likely to help generalize endoscopic hemostasis.

The current standard of endoscopic therapy consists of the use of hemoclips or thermo-coagulation with or without pre-injection with diluted epinephrine. TC-325 is a proprietary, inert inorganic mineral blend powder approved by FDA for the purpose of hemostasis. In the United States the powder is used for compression treatment of bleeding from external injuries in both civilian and combat casualties. The powder is highly absorbent. When in contact with fluid or blood the powder rapidly concentrates clotting factors at the bleeding site and forms an adherent coagulum. In 2011, Investigators reported the first endoscopic human application of the hemostatic powder TC-325. In 20 patients with Forrest type I bleeding from their gastro-duodenal ulcers, Investigators were able to control bleeding in 19 of them. The single patient with refractory bleeding from an angular gastric ulcer underwent angiography to his left gastric artery and a pseudo-aneurysm was found arising from the article. The aneurysm was successfully embolized with coils by angiographic methods. None of these patients needed surgery or died when followed up for 30 days. These initial results were encouraging. In gastroduodenal ulcers with Forrest I bleeding, rate of further bleeding would be around 55% if untreated by endoscopy.

Subsequent to this pilot study, several series were published on the endoscopic use of TC-325. The pooled rate in the initial control of bleeding with the use of TC-325 was 89.6%. Rate of further bleeding after hemostasis was 19.2%. The reported series consisted of patients with different case-mix but exclusively non-variceal in etiologies. Indications for use of TC-325 also varied in these series. The powder was used as mono-therapy, in combination to other endoscopic therapies or as a rescue therapy when conventional endoscopic treatment failed. In the absence of comparative studies, the role of TC-325 remains undefined.

Herein Investigators propose a randomized controlled study to compare endoscopic use of TC-325 as a mono-therapy to current standards of hemostasis using either hemo-clips or contact thermo-coagulation with or without diluted epinephrine in patients with active bleeding (Forrest type I) from non-variceal upper GI causes. Investigators hypothesize that endoscopic application of TC-325 would not be inferior in the control of bleeding from non-variceal sources when compared to standard treatment. If such is the case, endoscopic use of TC-325 may be preferred over existing techniques because of simplicity in TC-325 application. It appeals especially to endoscopists with less experience in endoscopic hemostasis. In lesions of challenging anatomical positions e.g. posterior bulbar duodenum, TC-325 may prove superior.

ELIGIBILITY:
Inclusion Criteria:

* patients with overt signs of upper gastrointestinal bleeding (hematemesis, melena and/or circulatory instability)
* documented bleeding (Forrest I) from a non-variceal upper gastrointestinal source (gastro-duodenal ulcers, Mallory Weiss tear, cancers, Dieulafoy's and other vascular lesions) at endoscopy.

Exclusion Criteria:

* without a full informed consent from the patient or his next of kin
* Age <18 years
* Pregnant
* Lactating women

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 224 (Actual)
Dates: Start 2015-09-07 (Actual); Primary Completion 2019-01-14 (Actual); Study Completion 2019-04-30 (Actual)

PRIMARY OUTCOMES:
number of participants who presents and confirmed endoscopically as recurrent upper gastro-intestinal bleeding | 30 days
  ( Further bleeding is defined by failure to control bleeding at index endoscopy, renewed hematemesis, fresh melena with circulatory instability after initial control of bleeding (systolic blood pressure of 90 mmHg or less or pulse rate of 110 per minute or more) and/or a drop in haemoglobin by 2 g/dl and haematocrit by 10% over 24 hours despite adequate transfusion. Further bleeding after initial endoscopic hemostasis requires documentation with immediate endoscopy which finds fresh blood and active bleeding from a previously treated upper GIB source. Patients with further bleeding after initial endoscopic control are considered to have reached an outcome endpoint.

SECONDARY OUTCOMES:
number of participants who required subsequent endoscopic treatment upon recurrent bleeding | 30 days
  number of participants who required subsequent endoscopic treatment upon recurrent bleeding
number of participants who required subsequent surgical treatment upon recurrent bleeding | 30 days
  number of participants who required subsequent surgical treatment upon recurrent bleeding
number of participants who required further blood transfusion post randomization | 30 days
  number of participants who required further blood transfusion post randomization
Days of hospitalization post randomization | 60 days
  Days of hospitalization post randomization
number of days which participant required caring in Intensive care unit post randomization | 60 days
  number of days which participant required caring in Intensive care unit post randomization
number of participants with adverse events as a Measure of Safety and Tolerability (related or unrelated to endoscopic treatment) | 30 days
  number of participants with adverse events as a Measure of Safety and Tolerability (related or unrelated to endoscopic treatment
number of participants with mortality from all causes within 30 days randomization. | 30 days
  number of participants with mortality from all causes within 30 days randomization
Ease of endoscopic treatment as measured by Visual Analog Scale reported by Endoscopist | 3 days
  self reported VAS scale: 0 cm to 10 cm
procedure time of endoscopic treatment | 3 days
  procedure time of endoscopic treatment
number of participant who need extra assistant to accomplish the endoscopic treatment | 3 days
  number of participant who need extra assistant eg advanced endoscopist to accomplish the endoscopic treatment other than the main endoscopist

CONTACTS AND LOCATIONS:
Overall Officials: JAMES YW LAU, MD, Principal Investigator — CUHK
Locations (1):
- Endoscopy Centre, Hong Kong, HONG KONG, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lau JYW, Pittayanon R, Kwek A, Tang RS, Chan H, Rerknimitr R, Lee J, Ang TL, Suen BY, Yu YY, Chan FKL, Sung JJY. Comparison of a Hemostatic Powder and Standard Treatment in the Control of Active Bleeding From Upper Nonvariceal Lesions : A Multicenter, Noninferiority, Randomized Trial. Ann Intern Med. 2022 Feb;175(2):171-178. doi: 10.7326/M21-0975. Epub 2021 Dec 7. PMID 34871051
- [Derived] Laine L, Barkun AN, Saltzman JR, Martel M, Leontiadis GI. ACG Clinical Guideline: Upper Gastrointestinal and Ulcer Bleeding. Am J Gastroenterol. 2021 May 1;116(5):899-917. doi: 10.14309/ajg.0000000000001245. PMID 33929377